CLINICAL TRIAL: NCT02219867
Title: Evaluation of Safety and Efficacy of Sub-anesthetic Ketamine Infusions as a Treatment for Patients Diagnosed With Resistant Major Depression
Brief Title: Ketamine Infusions for Major Depression Disorder
Acronym: Ketamie
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Revital Amiaz, Doctor, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sheba- Ketamine
Record Dates: First submitted 2014-08-12; First posted 2014-08-19 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Depressive Disorder, Major
Keywords: ketamine; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketamine (Experimental): Active Comparator
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Drug (including placebo)
  Other Names: ketalar

SUMMARY:
Ketamine has been safely used for induction and maintenance of anesthesia for decades and more recently has been used for chronic pain. Ketamine is a noncompetitive, high-affinity antagonist of the N-methyl-D-aspartate type glutamate receptor, with additional effects on dopamine and μ-opioid receptors. During the last 9 years several uncontrolled reports have been published, showing a rapid and impressive effect of ketamine in TRD patients (Berman, Cappiello et al. 2000; Zarate, Singh et al. 2006; Mathew, Murrough et al. 2010; Aan Het Rot, Zarate et al. 2012; Mathew, Shah et al. 2012; Murrough, Iosifescu et al. 2013). Recently three placebo-controlled trials showed that a single dose of sub-anesthetic, (0.5 mg/kg) slow intravenous (IV) ketamine improves depressive symptoms dramatically. Across studies, a clinically significant antidepressant response was maintained for up to 72 hours in 12 of 25 patients. Nonetheless, all but two patients relapsed <2 weeks post-ketamine (Zarate, Singh et al. 2006; aan Het Rot, Zarate et al. 2012). Rot et al. showed that repeated IV ketamine infusions prolongs the duration of improvement.

The investigators believe that the data presented above allows us to provide ketamine treatment here in the Sheba Medical Center for TRD patients.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is one of the leading causes of disability worldwide (Collins, Patel et al. 2011). A substantial proportion of patients do not achieve adequate remission despite multiple antidepressant trials and augmentation strategies (Rush, Trivedi et al. 2006; Weissman, Pilowsky et al. 2006). Treatment-resistant major depression (TRD) is defined as an insufficient response to at least two adequate antidepressant trials (Rush, Trivedi et al. 2006). Many of these patients are referred to previous somatic treatment e.g. electroconvulsive therapy (ECT), rapid Transcranial Magnetic Stimulation (rTMS) and Vagal Nerve Stimulation (VNS), all of which have serious disadvantages and/or limited efficacy.

Ketamine has been safely used for induction and maintenance of anesthesia for decades and more recently has been used for chronic pain. Ketamine is a noncompetitive, high-affinity antagonist of the N-methyl-D-aspartate type glutamate receptor, with additional effects on dopamine and μ-opioid receptors. During the last 9 years several uncontrolled reports have been published, showing a rapid and impressive effect of ketamine in TRD patients (Berman, Cappiello et al. 2000; Zarate, Singh et al. 2006; Mathew, Murrough et al. 2010; Aan Het Rot, Zarate et al. 2012; Mathew, Shah et al. 2012; Murrough, Iosifescu et al. 2013). Recently three placebo-controlled trials showed that a single dose of sub-anesthetic, (0.5 mg/kg) slow intravenous (IV) ketamine improves depressive symptoms dramatically. Across studies, a clinically significant antidepressant response was maintained for up to 72 hours in 12 of 25 patients. Nonetheless, all but two patients relapsed <2 weeks post-ketamine (Zarate, Singh et al. 2006; aan Het Rot, Zarate et al. 2012). Rot et al. showed that repeated IV ketamine infusions prolongs the duration of improvement.

The investigators believe that the data presented above allows us to provide ketamine treatment here in the Sheba Medical Center for TRD patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive disorder, chronic and/or recurrent of at least at moderate severity, determined as reflected by baseline scores of ≥32 on the Inventory of Depressive Symptomatology -Clinician rated IDS-C30
* Patients with demonstrated insufficient response to ≥2 adequate antidepressant trials in the current episode

Exclusion Criteria:

* Current psychotic or dissociative symptoms
* Severe personality disorder with psychosis or dissociative symptoms
* Lifetime history of psychotic mania
* Substance use disorder
* Current suicidal ideation
* Uncontrolled elevated blood pressure, non-sinus rhythm, unstable ischemic heart disease, uncorrected hyper thyroidism, and for women, pregnancy or the initiation of or female hormonal treatment <3 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-01 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Rating scale - MADRS | 24 hours after treatment

SECONDARY OUTCOMES:
Side effects monitoring | Up to 4 hours after ketamine infustion
  Blood pressure monitoring Dissociative symptoms detection and description

OTHER OUTCOMES:
Hamilston depression Rating Scale | Up to 30 days from last treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba MC, Ramat Gan, Israel